CLINICAL TRIAL: NCT05385432
Title: Induction in Sensitized Kidney Transplant Recipients Without Preexisting Donor-specific antiboDies: a Randomized Multicentre Trial Between a Lymphocyte Depleting and Basiliximab.
Brief Title: Induction in Sensitized Kidney Transplant Recipients Without Pre-existing Donor-specific antiboDies
Acronym: INSTEAD
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DR210298 - INSTEAD
Record Dates: First submitted 2022-03-04; First posted 2022-05-23 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-09

CONDITIONS: Renal Transplant Rejection; Induction Therapy
Keywords: Kidney transplantation; Basiliximab; ATG; induction; rejection
MeSH Terms: conditions — Rejection, Psychology | interventions — Antilymphocyte Serum; Mycophenolic Acid; Steroids; Basiliximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rabbit antithymocyte globulin (rATG) (Experimental): The infusion of rATG (Thymoglobulin® (1.5mg/kg/day, maximum daily dose: 100 mg)) starts just after the randomization pre-operatively on a functional arteriovenous fistula or a high-flow venous catheter during 3 to 7 days until efficient tacrolimus level is obtained. The recommended initial tacrolimus dose is Prograf® 0.1mg/kg/day twice day.
  Interventions: Drug: Rabbit Anti thymocyte globulin (rATG)
- Basiliximab (Active Comparator): The infusion of Basiliximab (Simulect® (20mg)) starts before the surgery on peripheral vein for 15 minutes and the second infusion at day 4.
  Interventions: Drug: Basiliximab

INTERVENTIONS:
Drug: Rabbit Anti thymocyte globulin (rATG) — The infusion of rTAG (Thymoglobulin® (1.5mg/kg/day, maximum daily dose: 100 mg)) starts just after the randomization pre-operatively on a functional arteriovenous fistula or a high-flow venous catheter during 3 to 7 days until efficient tacrolimus level is obtained.
  Other Names: Maintenance immunosuppressive regimen is the same in experimental and control groups combining tacrolimus, mycophenolate mofetil (MMF) or enteric-coated mycophenolate sodium (EC-MPS) and steroids
  Arms: rabbit antithymocyte globulin (rATG)
Drug: Basiliximab — Simulect® IV 40mg D0 and D4
  Other Names: Maintenance immunosuppressive regimen is the same in experimental and control groups combining tacrolimus, mycophenolate mofetil (MMF) or enteric-coated mycophenolate sodium (EC-MPS) and steroids
  Arms: Basiliximab

SUMMARY:
Induction therapy decreases the rate of acute allograft rejection in kidney transplant recipients (KTRs) and is strongly recommended. Polyclonal lymphocyte-depleting antibodies and interleukin-2 receptor (IL2R) antagonists are therefore widely used around the world, with a leading position for rabbit anti-thymocyte globulin (rATG, Thymoglobulin®) and basiliximab (Simulect®), respectively. The actual immunological risk of the sensitized KTRs without donor specific antibodies (DSAs) is still debated. The benefit-risk equation of lymphocyte depleting antibodies (versus IL2R antagonists) is not known in sensitized KTRs without DSAs. This clinical trial will compare the efficacy and safety of basiliximab and rATG in sensitized KTR without pre-existing DSAs detected by Luminex.

DETAILED DESCRIPTION:
Kidney transplantation is the first-line treatment of end stage renal disease, improving life expectancy and quality of life in comparison to dialysis. The success of transplantation is a consequence of major advances, especially the development of efficient immunosuppressive drugs. However, thousands of kidney transplants fail yearly around the world, and kidney allograft failure is known as an important case of end-stage renal disease, leading to increased morbidity, mortality and costs. To improve graft survival is therefore a priority, especially in a context of organ shortage.

Many risk factors of kidney graft loss have been identified but alloimmune response remains the first determinant of graft loss. This powerful donor specific immune response involves numerous effectors that may be harmful to the graft, such as T and B lymphocytes and antibodies. Those antibodies are mainly directed against human leucocyte antigens (HLA) and DSAs can be detected and identified in serum of sensitized KTRs. Alloreactivity T-cells and antibodies may induce distinct categories of acute and chronic graft damages. Lesions of rejection, recognized on tissue fragments sampling by percutaneous ultrasound-guided core needle graft biopsy, are classified and graded according to international Banff classification that is regularly updated. Two categories of biopsy-proven acute rejections (BPAR) are thus distinguished: T-cell mediated rejection (TCMR) and antibody-mediated rejection (ABMR). TCMR is a well-known risk factor of graft loss and also associated with subsequent de novo DSAs appearance. ABMR is considered as the first cause of kidney graft loss. In contrast to TCMR, that is usually sensitive to steroids, no treatment is able to completely block the production of DSA and reverse the process of ABMR, especially chronic ABMR. Prevent appearance of DSA and subsequent ABMR is therefore a major concern to improve kidney transplant outcome.

Appearance of DSA after transplantation (de novo DSA) depends mainly on number of HLA mismatches between donor and recipient and level of immunosuppression. Regarding immunosuppression, two clinical trials have reported an increased incidence of de novo DSA in patients receiving a calcineurin inhibitor-free maintenance treatment. In addition, some retrospective studies have suggested that mycophenolic acid would be more efficient to prevent de novo DSA formation. Standard-of-care for maintenance immunosuppression is therefore a combination of anticalcineurin (tacrolimus has widely replaced cyclosporin over last two decades), mycophenolic acid (mycophenolate mofetil or enteric-coated mycophenolate sodium) and steroids. Data about induction therapy (i.e. initial immunosuppressive treatment given during the first post-transplantation week) and risk of de novo DSA and ABMR are scarce.

Induction therapy is a pivotal component of the immunosuppressive treatment. It has decreased the rate of acute allograft rejection in KTRs and is strongly recommended. Polyclonal lymphocyte-depleting antibodies and interleukin-2 receptor (IL2R) antagonists are thus widely used around the world, with a leading position for rabbit anti-thymocyte globulin (rATG, Thymoglobulin®) and basiliximab (Simulect®), respectively. Today, these two induction treatments are used in common practice in kidney transplantation (rATG since 1984 and basiliximab since 2003). According to international KDIGO recommendations, IL2R antagonists are the first-line induction therapy in low-immunological risk no sensitized recipients (level 1, grade A), while immunosuppressive intensification using lymphocyte depletive agents is warranted in high-immunological KTRs (level 2, grade A). This intensification is supported by two randomized clinical trials that found rATG as more efficient to prevent acute rejection in recipients with a high immunological risk.

The current concern is that the definition of "immunological risk" used in those studies and international recommendations is no longer in line with current clinical practices. Indeed, immunological risk was estimated by the number of previous transplantations, recipient age, donor age, ethnicity, number of HLA mismatches and level of sensitization (calculated panel-reactive antibodies (cPRA) > 30%), based on cytotoxicity and ELISA techniques. Nowadays, highly sensitive single HLA-antigen flow bead (SAB) assays have replaced cytotoxicity and ELISA techniques in all French histocompatibility laboratories to detect low amounts of anti-HLA antibodies and accurately determine their specificity. It is therefore possible to characterize with a great precision whether a KTR is sensitized (i.e. presence of any anti-HLA antibody, irrespective of its specificity) and has anti-HLA antibody specific for DSA. Hence, the broad use of SAB assays has split sensitized KTRs in two distinct groups: those with at least one pre-transplant DSA, who have undoubtedly a high risk of BPAR and graft loss, and those without DSA. The actual immunological risk of the sensitized KTRs without DSA is still debated. Some studies have suggested that the presence of non-donor specific anti-HLA antibodies would represent an intermediate risk for graft loss and antibody mediated rejection and others that these antibodies did not affect graft outcome and risk of BPAR. A prospective study that compared rATG and basiliximab has recently confirmed that rATG should be used in sensitized KTRs with low amount of DSA detectable using SAB assay. Finally, the benefit-risk equation of lymphocyte depleting antibodies (versus IL2R antagonists) remains unknown only in sensitized KTRs without DSA.

Address this concern is very important because rATG has the potential to induce long lasting CD4+ T-cell depletion which may last for many months or even for many years. This prolonged CD4 T-cell lymphopenia has been shown to be associated with an increase of morbidity and mortality after renal transplantation. Indeed, profound CD4 T-cell lymphopenia (i.e. less than 200-/mm3) exposes to an increase of viral infection and rATG has been identified as a risk factor for BK virus (BKv) replication and cytomegalovirus (CMV) infection. The increase of the risk of post-transplant lymphoproliferative disorder and/or solid cancer in patients treated with rATG compared to the use of IL2R antagonists is still under debate. Because of the potential side effects related to rATG, the use of lymphocyte depleting agents should be limited only to patients who may benefit from its use compared to IL2R antagonists. Some kidney transplant centers have recently decided to use basiliximab instead of rATG in sensitized KTR without DSA before transplantation, in order to decrease the risk of infection and malignancies. Investigators puslished a monocentric case control study that suggested that basiliximab was associated with an unusual high risk of rejection and DSA appearance in this specific population. Similar alert regarding basiliximab has been recently reported in a small prospective study even though lack of power precludes any definitive conclusions. The prescription of induction treatment is currently heterogeneous according to the centers. These results highlight the urgent need of a new clinical trial to compare basiliximab and rATG in sensitized KTR without pre-existing DSAs.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18-79
* Registered on the transplant waiting list
* At least one anti-HLA antibody identified by the Luminex Single Antigen test with MFI ≥ 2000 (MFI threshold in agreement with French kidney allocation system.)
* Graft incompatibility rate (TGI) < 85%
* Ability for participant to comply with the requirements of the study
* Written informed consent obtained from the participant
* Participants covered by or entitled to social security.

Exclusion Criteria:

* DSA (negative virtual crossmatch with MFI threshold at 1000)
* Combined transplantation
* Usual contraindications to a kidney transplantation such as morbid obesity (BMI > 40 kg/m2), active drug abuse, uncontrolled psychiatric disease, or decompensated heart failure
* Beneficiaries of kidney transplants from donations after uncontrolled circulatory death (Maastricht II)
* Incompatible ABO transplantation
* Leukopenia lower than 3000/mm3
* Thrombocytopenia (platelets < 50G/L)
* Donor EBV Positive / Recipient EBV Negative
* Active HIV infection (positive viral charge)
* History of solid cancer (< 5 years), except to skin carcinoma (squamous-cell and basal-cell carcinoma).History of some solid cancer (prostate, breast) can be reduced (<2 years), depending on the prognosis for cancer recurrence as assessed by the oncologist.
* History of lymphoma
* Patients with severe uncontrolled systemic infection or severe allergy requiring acute or chronic treatment; Aspartate aminotransferase (ASAT), Alanine Amino Transferase (ALAT) or bilirubin greater than 3 times normal
* Known hypersensitivity or contra-indication to rabbit proteins, basiliximab including the product excipients
* Contra-indication to tacrolimus,mycophenolic acid ans steroids
* Pregnant or breastfeeding woman, or woman of childbearing potential not using a highly effective method of contraception, or having a desire to conceive, during the whole trial duration. A β-HCG test will be performed for inclusion.
* Patient under judicial protection, deprivation of liberty
* Participation in other interventional research with an investigational drug or medical device.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Estimated)
Dates: Start 2023-09-12 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2030-03-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of biopsy-proven acute rejection (BPAR) at year 1 | during the first post-transplantation year
  Incidence of BPAR (treated suspicious TCMR and confirmed TCMR with grade ≥ 1 and ABMR) in rATG and basiliximab groups, determined after blind central reading according to Banff 2019 classification.

SECONDARY OUTCOMES:
Incidence of BPAR in rATG and basiliximab groups at year 3. | at year 3
  Incidence of BPAR (suspicious and confirmed TCMR with grade ≥ 1 and ABMR) in rATG and basiliximab groups at year 3.
Incidence of composite criteria | at year 3
  Incidence of composite criteria including BPAR (suspicious and confirmed TCMR with grade ≥ 1 and ABMR), death and graft loss (retransplantation or dialysis) at year 3.
Incidence of confirmed TCMR and ABMR in rATG and basiliximab groups at year 1 and 3. | at year 1 and 3
  Incidence of confirmed TCMR and ABMR in rATG and basiliximab groups at year 1 and 3.
Incidence of de novo DSA in rATG and basiliximab groups at year 1 and 3 | at year 1 and 3
  Incidence of de novo DSA in rATG and basiliximab groups at year 1 and 3
Incidence of CMV viremia, CMV disease, BKv viremia and BKv nephropathy in rATG and basiliximab groups at year 1 and 3. | at year 1 and 3
  Incidence of CMV viremia, CMV disease, BKv viremia and BKv nephropathy in rATG and basiliximab groups at year 1 and 3.
Estimated glomerular filtration rate (eGFR) according to MDRD formula and proteinuria/creatinuria ratio in rATG and basiliximab groups at year 1 and 3 | at year 1 and 3
  Estimated glomerular filtration rate (eGFR) according to MDRD formula and proteinuria/creatinuria ratio in rATG and basiliximab groups at year 1 and 3
Incidence of primary and secondary outcomes (BPAR, TCMR, ABMR, death, graft loss, de novo DSA, CMV and BKv infections, eGFR) in subgroups defined by rank of transplantation. | at year 1 and 3
  ncidence of primary and secondary outcomes (BPAR, TCMR, ABMR, death, graft loss, de novo DSA, CMV and BKv infections, eGFR) in subgroups defined by rank of transplantation.
Health-Economics endpoints: Incremental Cost Utility Ratio | at year 1
  Incremental Cost Utility Ratio (ICUR) estimating the "cost per QALY gained", at 12 months, from the French Healthcare Insurance perspective, of rATG in comparison to basiliximab.
Health-Economics endpoints: Incremental Cost Effectiveness Ratio | at year 1
  Incremental Cost Effectiveness Ratio (ICER) estimating the "cost per prevented BPAR" at 12 months, from the French Healthcare Insurance perspective, of rATG in comparison to basiliximab.
Assessment of the safety | from date of randomization until the last visit at year 3 (the end of the follow-up for the patient)
  Assess the safety of rATG and basiliximab in sensitized kidney Transplant recipients without pre-existing donor-specific antibodies

REFERENCES:
- [Result] Goumard A, Sautenet B, Bailly E, Miquelestorena-Standley E, Proust B, Longuet H, Binet L, Baron C, Halimi JM, Buchler M, Gatault P. Increased risk of rejection after basiliximab induction in sensitized kidney transplant recipients without pre-existing donor-specific antibodies - a retrospective study. Transpl Int. 2019 Aug;32(8):820-830. doi: 10.1111/tri.13428. Epub 2019 Apr 12. PMID 30903722
- [Derived] Wajih Z, Karpe KM, Walters GD. Interventions for BK virus infection in kidney transplant recipients. Cochrane Database Syst Rev. 2024 Oct 9;10(10):CD013344. doi: 10.1002/14651858.CD013344.pub2. PMID 39382091